CLINICAL TRIAL: NCT00724425
Title: A Phase 1 Dose Escalation Study of the Safety and Pharmacokinetics of IPI-493 Orally Administered to Patients With Advanced Malignancies
Brief Title: A Phase 1 Dose Escalation Study of IPI-493
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug exposure of retaspimycin HCl was superior to IPI-493, Infinity will focus exclusively on retaspimycin
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-493-01
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Advanced Malignancies
MeSH Terms: interventions — tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: IPI-493 — Capsules, Multiple Schedules

SUMMARY:
IPI-493 is a potent inhibitor of heat shock protein 90 (Hsp90) and is orally bioavailable via a novel formulation.

DETAILED DESCRIPTION:
Hsp90 controls the proper folding, function, and stability of various "client" proteins within cells. Many of the clients of Hsp90 (such as Akt, Bcr-Abl, EGFR, Flt-3, c-Kit and PDGFR α) are oncoproteins or important cell-signaling proteins, and therefore are critical for tumor cell growth and survival. Inhibition of Hsp90 results in degradation of these proteins, which abrogates growth and survival signaling and leads to tumor cell death.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have pathologically confirmed advanced solid tumors
2. Progressive disease for their advanced solid tumor
3. Patients must be ≥18 years of age
4. Performance status of 0 or 1.
5. Not Pregnant by blood or urine test, and be willing to use adequate methods of birth control

Exclusion Criteria:

1. Treatment with the following therapies within the specified time period:

   * Any chemotherapy (other than nitrosoureas or mitomycin C), radiation therapy (other than whole brain irradiation [WBI]), surgery, hormonal therapy, or investigational therapy within 4 weeks of the start of IPI 493 administration
   * Any tyrosine kinase inhibitor (e.g., erlotinib, imatinib) within 2 weeks
   * Whole brain irradiation therapy within 3 months
   * Stereotactic cranial radiosurgery (SRS) within 4 weeks
   * Nitrosoureas or mitomycin C within 6 weeks
   * Any known Hsp90 inhibitor
2. Toxicities from prior therapies must have resolved to ≤ Grade 1 or baseline
3. Concurrent administration of the medications or foods , which are known to inhibit or induce CYP3A activity to a clinically relevant degree, is not allowed.
4. Concurrent treatment with any agent known to prolong the QTc interval
5. Known human immunodeficiency virus (HIV) positivity.
6. Inadequate hematologic function defined by absolute neutrophil count (ANC) < 1,500 cells/mm3, a platelet count < 100,000/mm3, and a hemoglobin < 9.0 g/dL
7. Inadequate hepatic function
8. Inadequate renal function
9. Sinus bradycardia
10. Baseline QTcF > 450 msec in males; QTcF > 470 msec in females.
11. Presence of left bundle branch block (LBBB), right bundle branch block (RBBB) if accompanied by left anterior hemiblock, bifascicular block or 3rd degree heart block. This does not include patients with a history of these events with adequate control by pacemaker.
12. Patients who have received > 450 mg/m2 of any anthracycline during prior chemotherapy must have a baseline left ventricular ejection fraction (LVEF) > 40%.
13. Active keratitis or keratoconjunctivitis.
14. Presence of active infection or systemic use of antibiotics within 72 hours of treatment.
15. Patients with a clinically active brain metastasis
16. Patients with a history of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months.
17. Significant co-morbid condition or disease which in the judgment of the Investigator would place the patient at undue risk or interfere with the study. Examples include, but are not limited to cirrhotic liver disease, sepsis, and other conditions.
18. Women who are pregnant or lactating.
19. Patients who have had a venous thromboembolic event (e.g., pulmonary embolism or deep vein thrombosis) requiring anticoagulation and meet any of the following criteria are excluded:

    * Have been on a stable dose of anticoagulation for <1 month
    * Have had a Grade 2, 3 or 4 hemorrhage in the past month
    * Are experiencing continued symptoms from their venous thromboembolic event

      * Patients who have had a venous thromboembolic event but do not meet any of the above three criteria are eligible for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To determine the safety and maximum tolerated dose (MTD) of IPI 493 | ongoing
To recommend a dosing regimen (dose and schedule) for subsequent studies of IPI 493 | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, MD, Study Director — Infinity Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - Premiere Oncology, Arizona, Scottsdale, Arizona
  - San Diego Pacific Oncology and Hematology Associates, Encinitas, California
  - Premiere Oncology, California, Santa Monica, California
  - Univeristy of Colorado Health Science Center, Aurora, Colorado
  - Mary Crowley Cancer Research Center, Dallas, Texas